CLINICAL TRIAL: NCT07267143
Title: Does a Highly Filled Injectable Resin Composite Work Better Alone or in Combination With a Nanohybride Resin Composite? A Randomised Clinical Trial
Brief Title: Does a Highly Filled Injectable Resin Composite Work Better Alone or in Combination With a Nanohybride Resin Composite?
Acronym: nanoinjectcomb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tolunay Aytas (Other)
Responsible Party: Sponsor-Investigator, Tolunay Aytas, research asistant in restorative dentistry, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/15-03
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Polydiastema Disorder
Keywords: High filled injectable composite polydiastema disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Injectable (Experimental): G-aenial Injectable (high filled injectable resin composite) group This study planned to investigate the clinical performance of G-aenial Injectable Universal (high filled ınjectable resin composite) in the treatment of anterior polydiastema disorders. This arm of the study is the group whose effectiveness was investigated. The results will be evaluated by comparing with a traditional anterior resin composite in terms of functional, biological and aesthetic properties.
  Interventions: Device: Highly Filled Injectable Composite (G-ænial Universal Injectable, GC Corp., Tokyo, Japan)
- Combine (Experimental): Restorations performed with a combined approach using a 1-mm palatal layer of nanohybrid composite resin (G-ænial A'Chord) followed by the injection of highly filled flowable composite resin (G-ænial Universal Injectable) guided by the PVS index.
  Interventions: Device: Nanohybrid Composite (G-ænial A'Chord, GC Corp., Tokyo, Japan); Device: Highly Filled Injectable Composite (G-ænial Universal Injectable, GC Corp., Tokyo, Japan)
- Conventional (Active Comparator): This group will serve as a "control". G-aenial Universal Injectable (high filled ınjectable resin composite) restorations will compare with the "G- Aenial A'chord" anterior resin composite restorations.
  Interventions: Device: Nanohybrid Composite (G-ænial A'Chord, GC Corp., Tokyo, Japan)

INTERVENTIONS:
Device: Nanohybrid Composite (G-ænial A'Chord, GC Corp., Tokyo, Japan) — Conventional nanohybrid resin composite (G-ænial A'Chord, GC Corp., Tokyo, Japan) was used for direct anterior veneer restorations. The material was applied using a free-hand layering technique following digital smile design and wax-up. A transparent silicone index (Exaclear, GC Corp.) was used for shape guidance when necessary. The enamel surfaces were etched with 37% phosphoric acid and bonded with a universal adhesive (G2 Bond, GC Corp.) before composite application. This intervention represents the standard clinical technique for direct composite veneers and serves as the active comparator group.
  Arms: Combine; Conventional
Device: Highly Filled Injectable Composite (G-ænial Universal Injectable, GC Corp., Tokyo, Japan) — Highly filled flowable injectable composite resin (G-ænial Universal Injectable, GC Corp., Tokyo, Japan) was used either as a sole restorative material or in combination with a nanohybrid composite for direct anterior veneers. For the injection process, a transparent PVS index (Exaclear, GC Corp.) was fabricated from a wax-up model and used to guide the placement of the material. In the combined technique, a 1-mm palatal layer of nanohybrid composite was placed first, followed by the injection of the flowable composite. The procedure aimed to improve adaptation, minimize voids, and optimize esthetic results compared to the conventional layering method.
  Arms: Combine; Injectable

SUMMARY:
This is a double blinded, randomized clinical study that evaluated the performance of a high filled injectable resin composite in polydiastema . The polydiastema disorders will be restored with high filled injectable resin composite (G'aenial Injectable Universal ) or anterior composite resin (G-aenial A'chord ). Restorations will be evaluated after 12 months according to FDI criteria and the data will be analyzed.

DETAILED DESCRIPTION:
: The aim of this study was to comparatively evaluate the clinical performance of a high filled injectable resin composite with an anterior composite resin (G-aenial A'chord) in polidaiastemas.

Participants who are 18 years of age or older and healthy, and who have applied to the Restorative Dentistry Department of Hacettepe University Faculty of Dentistry to receive treatment for polidiastema disorders on their front teeth will be included in the study. After explaining the purpose and conditions of the study, they will be asked to sign an informed consent form. The gender, age, and tooth numbers of the participants to be treated will be recorded. 240 upper incisors of 60 patients will be treated, with attention paid to the balanced distribution of teeth in the right and left arches...Data were will be analyzed with Chi- Square, Fisher's Exact Test, Mann U tests

ELIGIBILITY:
Inclusion Criteria:

* Polydiastema should be such that the mesial, distal and buccal surfaces of the tooth are included in the restoration.

  * 2. The patient has polydiastema in at least teeth 12, 11, 21 and 22
  * 3. The patient does not have a systemic disease that would prevent restorative treatment.
  * 4. The patient voluntarily signs the informed consent form
  * 5. The patient does not have a physical disability that may prevent him/her from coming for a check-up.
  * 6. The patient does not have a history of spontaneous pain in the teeth to be included.
  * 7. The patient's teeth are alive
  * 8. The patient does not have any periapical pathology in the relevant tooth.
  * 9. The patient's tooth to be included in the study must be in a position to be restored by direct method.
  * 10. The patient is between the ages of 18-35
  * 11. The patient has class 1 and class 2 bite

Exclusion Criteria:

* • 1.Participant must be under 18 years of age or over 35 years of age

  * 2. The participant has poor oral hygiene
  * 3. The participant has systemic disorders that may prevent regular attendance at treatment and control appointments.
  * 4. The participant has parafunctional habits such as clenching/grinding and biting foreign objects.
  * 5. Previous diastema closure or reshaping has been performed on the relevant teeth.
  * 6. Teeth whitening has been performed on the relevant teeth within the last week.
  * 6. Having severe periodontal problems in the relevant tooth
  * 7. The relevant tooth has previously been restored due to caries,
  * 8. The relevant tooth functions as a removable prosthesis support
  * 9. Teeth undergoing orthodontic treatment
  * 10. Finding the participant's breakeven and class 3 closure

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Functional properties score | 1 year
  The primary factor for determining the clinical performance of a restorative material is the Functional properties. Visual tactile examination tools will be used for evaluating restorations according to FDI criteria by two experienced researchers at 1- week 6-, 12- months. The functional properties are scored as 1- clinically excellent, 2- clinically good, 3-clinically sufficient/satisfactory, 4-clinically unsatisfactory 5-clinically poor (replacement necesessry). Clinically 1, 2 and 3 scores are clinical acceptable but 4 and 5 scores are designated as failure.
  [Time Frame: 1 year]
Esthetic properties score | 1 year
  The secondary factor for determining the clinical performance of a restorative material is the Esthetic properties. Visual examination will be used for evaluating restorations according to FDI criteria by two experienced researchers at 1- week 6-, 12-months. The Esthetic properties are scored as 1- clinically excellent, 2-clinically good, 3-clinically sufficient/satisfactory, 4-clinically unsatisfactory 5-clinically poor (replacement necesessry). Clinically 1, 2 and 3 scores are clinical acceptable but 4 and 5 scores are designated as failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No